CLINICAL TRIAL: NCT00453375
Title: A Randomized, Blinded, Placebo Controlled, Safety and Pharmacodynamic Study of BHT-3021 With Open Label Cross-Over in Subjects With Type I Diabetes Mellitus
Brief Title: Phase 1 Study of BHT-3021 in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayhill Therapeutics (Industry)
Responsible Party: Diane Amend, Clinical Trials Manager, Bayhill Therapeutics
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BHT-3021-01
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Hypoglycemia
Keywords: Diabetic; Diabetes; Type 1 Diabetes; Type 1 Diabetes Mellitus; autoimmune disease
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): BHT-3021
  Interventions: Drug: BHT-3021
- 2 (Placebo Comparator): BHT-Placebo
  Interventions: Drug: BHT-Placebo

INTERVENTIONS:
Drug: BHT-3021 — Evaluation of up to four dose levels will be given in weekly IM injections for 12 weeks.
  Arms: 1
Drug: BHT-Placebo — Evaluation of up to four dose levels will be given in weekly IM injections for 12 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety of BHT-3021 injections given weekly for 12 weeks and to evaluate the effect of BHT-3021 on antibody and immune (T cell) responses to autoantigens (e.g. insulin). Changes in pancreatic beta cell function, insulin requirements and blood glucose levels will also be evaluated.

DETAILED DESCRIPTION:
Type 1 diabetes results from an attack by the body's own immune system on the insulin producing cells in the pancreas. Around 80% of diagnosed patients have detectable antibodies to islet cell self-proteins including, insulin IA-2 and glutamic acid decarboxylase. The drug, BHT-3021 is being studied because an agent that stops autoimmune damage could offer patients benefit.

Study Description: A Randomized, Blinded, Placebo Controlled, Safety and Pharmacodynamic Study of BHT-3021 with Open Label Cross-Over in Subjects with Type I Diabetes Mellitus that will enroll up to 72 subjects in this trial. Subjects will be randomized to BHT-3021 or BHT-placebo in a 2:1 ratio.

The duration of the study is approximately 25 to 37 months depending on treatment assignment: 4 week Screening Period; 12 month Blinded Treatment and Evaluation Period; 12 month Cross-over Treatment and Evaluation Period (BHT-placebo subjects only); 12 month Long Term Follow-Up period.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Type 1a Diabetes Mellitus based on ADA Criteria
* ≤5 years since T1D was diagnosed
* ≥ 18 years of age
* ≤ 40 years of age at the time of diagnosis of Type 1a diabetes
* Presence of antibodies to at least one of the following antigens:

insulin, GAD-65, or IA-2

* Detectable fasting C-peptide level
* C-peptide increase during screening mixed meal tolerance test with a minimal stimulated value of ≥ 0.2 pmol/mL
* Presence of antibodies to at least one of the following antigens: insulin, GAD-65, or IA-2. If insulin antibody positive only, determination must be within 2 weeks of insulin initiation

Exclusion Criteria:

* BMI > 30 kg/m2
* Unstable blood sugar control defined as one or more episodes of severe hypoglycemia (defined as hypoglycemia that required the assistance of another person) within the last 30 days
* Current use of inhalable insulin
* Previous immunotherapy for T1D
* Administration of an experimental agent for T1D at any time or use of an experimental device for T1D within 30 days prior to screening, unless approved by the medical monitor
* History of any organ transplant, including islet cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this study is safety.Safety parameters include: stimulated C-peptide response levels, opthalmologic examination, laboratory assessments, 24-hr urine protein, allergic reactions and adverse events including hypoglycemia.

SECONDARY OUTCOMES:
The secondary endpoints are pharmacodynamic parameters. Parameters include plasmid levels and insulin mRNA levels in blood and urine, Stimulated C-peptide response and Immunological response.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gottlieb, MD, Study Chair — University of Colorado, Denver; Joanne Quan, MD, Study Director — Bayhill Therapeutics Inc.; Len Harrison, MD, Study Chair — Walter and Eliza Hall Institute of Medical Research
Locations (18):
- United States (10):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Valley Research, Fresno, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Private Practice, Denver, Colorado
  - MedStar Research Institute, Washington D.C., District of Columbia
  - University of Miami, Miller School of Medicine, Diabetes Research Institute, Miami, Florida
  - Private Practice, Wellington, Florida
  - Creighton Diabetes Center, Omaha, Nebraska
  - Diabetes and Glandular Disease Center, San Antonio, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- Australia (4):
  - Peninsula Clinical Research Centre, Kippa-Ring, Queensland
  - Royal Melbourne Hospital, Parkville, Victoria
  - Eastern Clinical Research Unit, Ringwood East, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- New Zealand (4):
  - Middlemore Hospital, Otahuhu, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Regional Diabetes Service, Hamilton, Waikato Region
  - The Diabetes Centre, Newtown, Wellington Region

REFERENCES:
- See also: Bayhill Therapeutics Inc., Click Here for More Information Regarding this Study. — http://www.bayhilltx.com